CLINICAL TRIAL: NCT02345785
Title: Evaluation of the Change of Penile Corpus Cavernosum After Caudal Block Using Ultrasonography in Children
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0891
Record Dates: First submitted 2015-01-12; First posted 2015-01-26 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Pediatric Urologic Surgeries
MeSH Terms: interventions — Urologic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: pediatric patients who need urologic surgery and caudal block
  Interventions: Other: urologic surgery and caudal block

INTERVENTIONS:
Other: urologic surgery and caudal block

SUMMARY:
The purpose of this study is to evaluate the change of penile corpus cavernosum after caudal block using ultrasonography in pediatric patient.

ELIGIBILITY:
Inclusion Criteria:

1. Twenty (ASA status I or II) children, ages 2 to 7 yr old, who were scheduled for a urologic surgery
2. Children who needed caudal block for postoperative analgesia

Exclusion Criteria:

1. if there were contraindications for caudal block including hypersensitivity to any local anaesthetics, bleeding diathesis, infections at the puncture sites, or pre-existing neurological disease.
2. patients scheduled for penile surgery

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients who need urologic surgery and caudal block
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-10-02; Primary Completion 2016-01-22 (Actual); Study Completion 2016-01-22 (Actual)

PRIMARY OUTCOMES:
change of penile corpus cavernosum | 1 min after LMA insertion
  Evaluation of the change of penile corpus cavernosum after caudal block using ultrasonography in children
change of penile corpus cavernosum | 2 min after caudal block
  Evaluation of the change of penile corpus cavernosum after caudal block using ultrasonography in children
change of penile corpus cavernosum | 5 min after caudal block
  Evaluation of the change of penile corpus cavernosum after caudal block using ultrasonography in children

SECONDARY OUTCOMES:
cavernosal arterial hemodynamics | 1 min after LMA insertion
  Investigation of cavernosal arterial hemodynamics included peak systolic velocity [PS], end diastolic velocity [ED], mean velocity [MV], time-averaged maximum velocity [TAmax], time-averaged mean velocity [TAmean], pulsatility index [PI], volume flow [VF], and dorsalis pedis artery diameter [D].
cavernosal arterial hemodynamics | 2 min after caudal block
  Investigation of cavernosal arterial hemodynamics included peak systolic velocity [PS], end diastolic velocity [ED], mean velocity [MV], time-averaged maximum velocity [TAmax], time-averaged mean velocity [TAmean], pulsatility index [PI], volume flow [VF], and dorsalis pedis artery diameter [D].
cavernosal arterial hemodynamics | 5 min after caudal block
  Investigation of cavernosal arterial hemodynamics included peak systolic velocity [PS], end diastolic velocity [ED], mean velocity [MV], time-averaged maximum velocity [TAmax], time-averaged mean velocity [TAmean], pulsatility index [PI], volume flow [VF], and dorsalis pedis artery diameter [D].

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea